CLINICAL TRIAL: NCT03533426
Title: The Impact of Ultrasound-guided Serratus Anterior Plane Catheter Block (SAPB) Following Thoracotomy for Chest Malignancies on the Emergence of Post-thoracotomy Pain Syndrome (PTPS): A Pilot Study
Brief Title: Ultrasound-guided Serratus Block and the Emergence of Post-thoracotomy Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ehab Hanafy Shaker, Principal investigator, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Raafat-Ehab.serratus
Record Dates: First submitted 2018-04-23; First posted 2018-05-23 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Thoracic Neuritis
MeSH Terms: interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the data collector will be blinded to the study groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pump based patient controlled analgesia (Active Comparator): Analgesia is maintained using disposable silicon ballon pump "Accufuser" containing morphine 0.2 mg/ml, 8mg ondansetron plus and 180 mg ketorolac. The infusion rate is 5 ml / h and lockout interval of 15min. the hourly delivered morphine dose is 1-1.8 mg & the pump is sufficient for about 60 hours according to patient response.
  Interventions: Procedure: Patient controlled analgesia
- serratus anterior plane catheter block (Active Comparator): Linear ultrasound transducer (superficial) 6-12 MHz is utilized to count the ribs up to 4th or 5 th rib in the mid-axillary line. Musculature of thoracic wall is identified sonographically,an echogenic needle "14-16 G, 100 mm" is inserted in plane with the U/S probe towards the plane deep to the serratus anterior muscle. Under real - time U/S, single shot of 20ml contrast medium "iohexol = omnipaque" 150 mg I2 / ml is injected to check the plane and level (T3-T8/9) of SAPB.A reinforced radiopaque catheter is threaded through the needle and its final position underneath the plane of serratus anterior muscle is confirmed fluoroscopically. 20ml 0.25% levobupivacaine (Chirocaine).Analgesia is maintained using 0.125% levobupivacaine infusion at a rate of 7-12 ml/h according to patient response.
  Interventions: Procedure: Serratus anterior plane catheter block

INTERVENTIONS:
Procedure: Serratus anterior plane catheter block — Ultrasonographic guided placement of a catheter under the serratus anterior muscle in cases of open thoracotomies for chest malignancies in an attempt to reduce the emergence of postthoracotomy pain syndrome.
  Arms: serratus anterior plane catheter block
Procedure: Patient controlled analgesia — The use of patient controlled analgesia through a pump aiming to reduce the development of postthoracotomy pain syndrome
  Arms: Pump based patient controlled analgesia

SUMMARY:
The aim of this prospective, single blinded, comparative pilot study is to evaluate U/S guided serratus anterior plane catheter block (SAPB) versus patient-controlled analgesia (PCA) on the emergence of post - thoracotomy pain syndrome (PTPS). The investigator's assumed hypothesis is that; SAPB is an effective thoracic analgesic technique that may reduce the development of PTPS.

DETAILED DESCRIPTION:
Lung cancer has the highest incidence of all malignancies worldwide & represents about 13% of all cancer victims. Lung cancer still represents the first cause of cancer deaths and lung resection surgeries could be the main therapeutic procedure. Hence, the number of thoracotomies is progressively increasing with more & more post- thoracotomy pain . Together with amputation, thoracotomy is considered the main etiology of severe & long-term acute and chronic post-surgical pain syndromes (CPSP). The prevalence of post - thoracotomy pain syndrome (PTPS) is variable (30-50%). The international association for the study of pain (IASP) has defined PTPS as "pain that recurs or persists along the thoracotomy scar at least 2 months after the procedure".Besides, PTPS is mostly described with neuropathic manifestations along the thoracotomy scar, mammary & submammary ipsilateral scapular & interscapular areas. Pain is often aching, burning with tingling, numbness, pruritis plus sensory loss and/or hypoesthesia.Preemptive post-thoracotomy analgesia is mostly multimodal & integrates both systemic & regional techniques. Systemic drugs (either given parenterally or through patient controlled - analgesia "PCA") include, NSAIDs, Cox - II inhibitors, paracetamol, opioids, ketamine (as N-methyl-D- aspartate blocker), gabapentins & pregabalin, selective serotonin re-uptake inhibitors and/or duloxetine .Regional analgesic techniques include thoracic epidural analgesia (TEA) which, is considered by many as the gold standard analgesic mode for post-thoracotomy pain .Other regional analgesic techniques are paravertebral analgesia (PVB), intercostal nerve blocks and intrapleural analgesia.Recently SAPB has been practiced more widely as an U/S - guided, simple technique of effective post-thoracotomy analgesia which is comparable with standard techniques such as TEA and PVB.

ELIGIBILITY:
Inclusion Criteria:

* age > 18y
* American Society of Anesthethiologists (ASA) physical status II or III .
* Patient will undergo thoracotomy for lung resection procedures (metastatectomy, segmentectomy lobectomy, pneumonectomy or pleuropneumonectomy).

Exclusion Criteria:

* Patients with history of drugs (opioids, L.A., NSAIDs) allergy.
* Morbid obese patients (BMI >40) .
* Major cardiorespiratory, hepatic, renal, endocrinal or hematological disorders.
* Patients on chronic analgesic therapy (daily morphine ≥ 30 mg or equivalent dose of other opioids).
* History of drug abuse and neuropsychiatric diseases .
* History of thoracic cancer surgery within the last five years or patients having chest recurrence within 6 months.
* Patients having severe intra or post-operative bleeding or demanding postoperative ventilation will be also excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Assessment for the possible emergence of post - thoracotomy pain syndrome . | changes in 4 and 12 weeks .
  The neuropathic PTPS cases are screened using the grading system for neuropathic pain (GSNP). Positive cases of PTPS having neuropathic component is grade 3 (probable) or 4 (definite) i.e GSNP ≥3 .

SECONDARY OUTCOMES:
Assessment of patient daily activity and functional capacity. | changes in 4 and 12 weeks .
  Activity of daily living score (ADL score).It comprises 6 basic daily activities (feeding, toilet, bathing, dressing, grooming and walking) with each item is scored either 1= need no help, 2=need some help, 3=need complete help
Assessment of patient's quality of life. | changes in 4 and 12 weeks .
  Flanagan quality of life scale.A 16 items (domains) questionnaire with each item weights 1 to 7 points.the total score ranges from 16 to 112 .Higher values indicate better quality of life .It will be explained to the patients by the pain physician and the total score will be calculated and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ehab H Shaker, MD, Principal Investigator — National Cancer Institute- Cairo University
Locations (1):
- Department of Anesthesia and Pain medicine.National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
the final results and conclusion can be shared after finishing and submitting the trial .

REFERENCES:
- See also: preventing and treating pain after thoracic surgery — http://anesthesiology.pubs.asahq.org/article.aspx?articleid=1923467